CLINICAL TRIAL: NCT06000332
Title: Evaluation of POC Pulse-dose Demand Oxygen Delivery for Nocturnal Hypoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INO-05
Record Dates: First submitted 2023-07-13; First posted 2023-08-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Nocturnal Hypoxemia
Keywords: hypoxemia, oxygen
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- InogenOne Rove 6 Portable Oxygen Concentrator (Experimental): InogenOne Rove 6 Portable Oxygen Concentrator
  Interventions: Device: InogenOne Rove 6 Portable Oxygen Concentrator

INTERVENTIONS:
Device: InogenOne Rove 6 Portable Oxygen Concentrator — overnight use of Portable Oxygen Concentrator, 6 hours minimum

SUMMARY:
The aim of this study is to describe the effect of the Inogen Rove 6 Portable Oxygen Concentrator on peripheral oxygen saturation in adults receiving supplemental oxygen at night and examine whether the device can adequately maintain oxygen saturation during sleep.

DETAILED DESCRIPTION:
The study design is a prospective, single site, single arm, open label, pilot study. The aim of this study is to describe the effect of the Inogen Rove 6 Portable Oxygen Concentrator on peripheral oxygen saturation in adults receiving supplemental oxygen at night and examine whether the device can adequately maintain oxygen saturation during sleep, i.e., achieve target with initial titration setting and/or with any needed adjustments of setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be of any gender
2. Subject's age must be 40 - 80 years
3. Subjects must have a current prescription for nocturnal oxygen < 3 L/min continuous or current use of a Portable Oxygen Concentrator.

Exclusion Criteria:

1. Subject is using any ancillary medical device(s) that may interfere with the operation of or data interpretation from the InogenOne device (such as CPAP/BiPAP, NIV).
2. Subjects with nasal obstruction
3. Subjects taking any drugs that affect respiratory center drive
4. Subject has an acute illness or hospitalization within the last 30 days
5. Subject has a change in medication within the last 15 days
6. Subject is currently receiving respiratory stimulant medications (such as acetazolamide, medroxyprogesterone, doxapram, theophylline/aminophylline, protriptyline and buspirone)
7. Subject has significant comorbidities that in the opinion of the Investigator would interfere with outcomes and/or study conduct
8. Subject's prescribed treatment is in conflict with study procedures
9. Subjects with any unstable disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Number/% of subjects that could achieve SpO2 ≥90% for >30% of sleep time | 6 hours overnight
  oxygen saturation (SpO2)

SECONDARY OUTCOMES:
Number/% of subjects requiring increased settings and the difference between initial and maximal settings required to meet target SpO2 ≥90% for >30% of sleep time criteria | 6 hours overnight
  oxygen saturation (SpO2)
Time/% time above/below 90% target on initial setting and maximal setting | 6 hours overnight
  oxygen saturation (SpO2)
Number, duration, variability, and AUC of dips below 90% during sleep time on initial setting and maximal setting | 6 hours overnight
  oxygen saturation (SpO2)
Minimum/maximum SpO2 on initial setting and maximal setting | 6 hours overnight
  oxygen saturation (SpO2)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Glezer, MD, Study Chair — Inogen Inc.
Locations (1):
- Piedmont Healthcare, Statesville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No